CLINICAL TRIAL: NCT02791646
Title: Optimizing Delivery of a Behavioral Cancer Pain Intervention Using a SMART
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00070823
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: PCST-Full (Pain Coping Skills Training); PCST-Brief

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCST-Full (Experimental): PCST-full will consist of a 5-session intervention delivered to participants at the medical center by their therapist.
  Interventions: Behavioral: Pain Coping Skills Training Full
- PCST-Brief (Experimental): Pain coping skills training brief (PCST-Brief) will consist of a 60 minute, in-person session followed by 4-weeks of daily text messaging
  Interventions: Behavioral: Pain Coping Skills Brief

INTERVENTIONS:
Behavioral: Pain Coping Skills Training Full — Pain Coping Skills Training Full(PCST-Full) will consist of a 5-session intervention delivered to participants at the medical center by their therapist.
  Arms: PCST-Full
Behavioral: Pain Coping Skills Brief — Pain coping skills training brief (PCST-Brief) will consist of a 60 minute, in-person session followed by 4-weeks of daily text messaging
  Arms: PCST-Brief

SUMMARY:
This trial is a sequential multiple assignment randomized trial (SMART), that will examine response to differing doses of a behavioral cancer pain intervention (Pain Coping Skills Training [PCST]) and subsequent response-based adjustments to doses. Cancer patients with pain will initially be randomized to receive either PCST-Full or PCST-Brief. Participants who do not report pain reduction to their initially assigned intervention will be re-randomized to receive either maintenance or an increased level of intervention. Participants who report pain reduction to their initially assigned intervention will be re-randomized to either a maintenance dose or no further treatment. Intervention responses will be compared across conditions using a standard two-sided, two-sample t-test. Techniques typically used for SMART studies will be used to compare intervention dosage sequences across PCTS that adjusts to initial dosage based on patient responses. The risk and safety issues in this trial are low and limited to those common to a psychosocial intervention (e.g., loss of confidentiality).

DETAILED DESCRIPTION:
The incidence of moderate to severe pain in cancer patients remains greater than 50%. NIH guidelines recommend the implementation of behavioral cancer pain interventions into patient care. Yet, implementation remains low. Evidence on patient dose-response (i.e., number of sessions, skills), intervention adaption based on initial response, and understanding personal characteristics related to differing dose-response can improve implementation by optimizing behavioral intervention delivery.

This trial is a sequential multiple assignment randomized trial (SMART), that will examine response to differing doses of a behavioral cancer pain intervention (Pain Coping Skills Training [PCST]) and subsequent response-based adjustments to doses. Cancer patients with pain (N=327) will initially be randomized to receive either PCST-Full or PCST-Brief. Participants who do not respond (<30% pain reduction) to their initially assigned intervention will be re-randomized to receive either maintenance (i.e., booster sessions focused on problem solving and skills reinforcement) or an increased level of intervention (i.e., additional sessions and skills). Participants who respond (> 30% pain reduction) to their initially assigned intervention will be re-randomized to either a maintenance dose or no further treatment. Intervention responses will be (% reduction in pain) will be compared across conditions using a standard two-sided, two-sample t-test. Techniques typically used for SMART studies will be used to compare intervention dosage sequences across PCTS that adjusts to initial dosage based on patient responses. The risk and safety issues in this trial are low and limited to those common to a psychosocial intervention (e.g., loss of confidentiality).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer (initial or recurrence) within the last two years
* being >18 years old
* having a life expectancy of at least 12 months
* having a pain intensity rating of >5.

Exclusion Criteria:

* cognitive impairment
* metastases to the brain
* presence of a severe psychiatric condition (i.e., psychotic disorder or episode) or a psychiatric condition (e.g., suicidal intent) that would contraindicate safe participation in the study as indicated by the medical chart, treating oncologist, or interactions with the medical/study staff
* current or past (<6 months) engagement in PCST for cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity | baseline to 6 weeks
  Pain intensity will be assessed by asking patients about their pain at its "worst", "least", "average", and "now". Patients will answer on a scale where 0 = "no pain" to 10 = "pain as bad as you can imagine". The worst, least, and average items will be asked in reference to the last 7 days. A composite averaged score of these four items will be used to represent pain intensity.
Change in Pain Intensity | Baseline, 6 weeks, 3 months and 6 months
  Pain intensity will be assessed by asking patients about their pain at its "worst", "least", "average", and "now". Patients will answer on a scale where 0 = "no pain" to 10 = "pain as bad as you can imagine". The worst, least, and average items will be asked in reference to the last 7 days. A composite averaged score of these four items will be used to represent pain intensity.

SECONDARY OUTCOMES:
Pain Interference | Baseline, 6 weeks, 3 months and 6 months
  Pain interference will be assessed with the Brief Pain Inventory (BPI). Pain interference will be assessed by asking patients how much their pain has interfered with seven daily activities including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep within the last 7 days. Answers will be on a 0 = "does not interfere" to 10 = "completely interferes" scale; items will be averaged to represent pain interference. These measures have been recommended for use in chronic-pain clinical trials.
Practicality as measured by accrual | 8 months
  Accrual will be indicated by meeting the recruitment goal of 327 participants during the proposed 48 months of recruitment (~7 participants per month)
Practicality as measured by retention | 8 months
  Retention will be indicated by 80% of consented participants completing the study protocol (i.e., remain enrolled)
Practicality as measured by adherence | 8 months
  Adherence for patients who are accrued to the study will be examined by calculating the proportion successfully completing all intervention sessions during their first randomization and second randomization
Pain Catastrophizing, as measured by the 6-item pain catastrophizing subscale of the Coping Strategies Questionnaire | Baseline, 6 weeks, 3 months and 6 months
  These items ask about patients tendency to catastrophizing when faced with pain (e.g., "When I feel pain it is awful and it overwhelms me") and are answered on a 0 = never to 6 = always scale. Items are summed for a total score
Cost-Effectiveness | 8 months
  We will create a composite cost variable based on patient time, provider time, and the EQ-5D.The EQ-5D is a measure of health status that can be linked to population-based preference weights is widely used in economic evaluations. It is short, assessing 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The respondent indicates no problems, some problems, or severe problems in each dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara J Somers, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Li Y, Reed SD, Winger JG, Hyland KA, Fisher HM, Kelleher SA, Miller SN, Davidian M, Laber EB, Keefe FJ, Somers TJ. Cost-Effectiveness Analysis Evaluating Delivery Strategies for Pain Coping Skills Training in Women With Breast Cancer. J Pain. 2023 Sep;24(9):1712-1720. doi: 10.1016/j.jpain.2023.05.004. Epub 2023 May 13. PMID 37187219
- [Derived] Kelleher SA, Dorfman CS, Plumb Vilardaga JC, Majestic C, Winger J, Gandhi V, Nunez C, Van Denburg A, Shelby RA, Reed SD, Murphy S, Davidian M, Laber EB, Kimmick GG, Westbrook KW, Abernethy AP, Somers TJ. Optimizing delivery of a behavioral pain intervention in cancer patients using a sequential multiple assignment randomized trial SMART. Contemp Clin Trials. 2017 Jun;57:51-57. doi: 10.1016/j.cct.2017.04.001. Epub 2017 Apr 11. PMID 28408335